CLINICAL TRIAL: NCT01215162
Title: Phase II Study of Intra-Operative Electron Irradiation and External Beam Irradiation After Lumpectomy in Patients With T1N0M0 and T2N0M0 Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: William Wong M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1681-02; MCS066
Record Dates: First submitted 2009-08-07; First posted 2010-10-06 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Experimental): Patients with stage T1/T2No breast cancer receiving breast conserving treatment
  Interventions: Radiation: Intra-operative radiation to tumor bed

INTERVENTIONS:
Radiation: Intra-operative radiation to tumor bed — IOERT is given to the tumor bed. Applicator selection should allow treatment of the tumor bed plus 1-2 cm margin. The surgical incision may need to be enlarged slightly to allow the placement of the appropriate applicator. The use of more than 1 treatment field is discouraged. In order to encompass the entire tumor bed in 1 treatment field, it may be necessary to suture the mammary parenchyma loosely so that the lateral margins of the tumor bed are brought into apposition. Electron energy used for the treatment. If the tumor bed can be flattened and encompassed by an applicator, 6 MeV electron is recommended. Use of bolus material may be considered to increase the surface dose. If the mammary parenchyma has been brought into apposition by sutures, a higher electron energy may be necessary to allow adequate dose coverage to a depth of 1.0-2.0 cm into the tumor bed. The dose of IOERT is 1000 cGy, prescribed to the 90% isodose line.

SUMMARY:
The study is being done to determine the tolerance to single fraction intra-operative electron irradiation (IOERT) and external beam photon irradiation (EBRT) following lumpectomy for T1/T2N0M0 breast cancer. IOERT is used in lieu of the 5-8 days of electron beam boost irradiation that is usually given after EBRT. Data from two centers as well as preliminary data from a randomized trial in Europe suggest that IOERT boost is well tolerated and efficacious. In our study, patients will undergo standard lumpectomy and sentinel lymph node sampling or axillary dissection. After the lumpectomy, IOERT of 10 Gy will be delivered in a single fraction to the tumor bed by a mobile electron machine in the operating room. EBRT to the whole breast will be administered once the surgical wound has healed adequately. The primary objective is to determine the feasibility and acute patient tolerance to IOERT and EBRT after lumpectomy. Secondary objectives include assessment of local control and distant control of disease, as well as evaluation of long-term side effects and cosmetic outcome of the treatment.

ELIGIBILITY:
Eligibility:

1. Histologically proven primary invasive breast carcinoma.
2. Tumor pathologically determined <= 5cm in diameter.
3. Single, discrete, well-defined primary tumor.
4. Any micro-calcifications must be focal. A specimen radiograph is required after lumpectomy to assure removal of all malignant appearing calcifications.
5. Pathologically negative surgical margins.
6. Axillary lymph node status can be determined by level I and II lymph node dissection or sentinel lymph node sampling.
7. ECOG performance status 0-2.

Contraindications:

1. Multicentric disease and/or diffuse malignant appearing microcalcifications.
2. Evidence of metastatic breast cancer.
3. Axillary lymph node involvement.
4. Pre-existing collagen vascular disease except rheumatoid arthritis that does not require immunosuppressive therapy.
5. Prior irradiation to the ara of planned radiation field.
6. Pregnant or lactating women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2003-01; Primary Completion 2005-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility and acute patient tolerance of IOERT and EBRT after lumpectomy for patients with stage T1/T2N0M0 breast cancer. | weekly evaluation during 5 weeks of radiation
  To determine the acute skin reaction, breast edema, pnemonitis, cardiac side effects during radiation using RTOG acute toxicity scale
Determine the local tumor control and distant tumor control rates for patients with stage T1/T2N0M0 breast cancer. | every 6 months follow-up for 5 years, then yearly to end in 04/2013
Determine long-term side effects and cosmetic outcome of IOERT to tumor bed and EBRT after lumpectomy for patients with stage T1/T2N0Mo breast cancer. | every 6 months follow-up for 5 years, then yearly to end in 04/2013
  To determine the late skin reaction, breast edema, pneumonitis, cardiac side effects during radiation using RTOG late toxicity scale

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States